CLINICAL TRIAL: NCT04598061
Title: IV Dexmedetomidine as Spinal Anesthesia Adjuvant in Infants : RACHI_dex
Brief Title: IV Dexmedetomidine as Spinal Anesthesia Adjuvant in Infants
Acronym: RACHI_dex
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0521
Record Dates: First submitted 2020-10-06; First posted 2020-10-22 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Newborns; Infant; Spinal Anesthesia
Keywords: less than 7 kg; undergoing an infra-umbilical surgery; Spinal anesthesia; Dexmedetomidine; respiratory complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Newborns or Infants less than 7 kg undergoing an infra-umbilical surgery: Newborns or Infants less than 7 kg undergoing an infra-umbilical surgery
  Interventions: Drug: Dexmedetomidine IV

INTERVENTIONS:
Drug: Dexmedetomidine IV — Dexmedetomidine IV

SUMMARY:
* Spinal anesthesia in newborns is one of " Gold standard " techniques in short subumbilical surgeries (less than 30 minutes) with advantage of avoiding the risks inherent to general anesthesia.
* Spinal anesthesia of the newborn remains a complex technical procedure with a failure rate of up to 16%. The child's movements and certain degrees of discomfort may also interfere with the successful completion of the procedure.
* The second major issue of spinal anesthesia is the limitation of the motor block duration and the need for general anesthesia to complete the surgery
* Spinal anesthesia duration can be prolonged by the addition of differents adjuvant such as opioid or alpha 2 adrenergic agonist.
* Since 2018, dexmedetomidine, an alpha 2 adrenergic agonist with sedative, analgesic and anxiolytic properties, is being used as a current and standard practice in our anesthesia department. Intravenous administrationis performed ten to twenty minutes before spinal anesthesia placement in all children weighing less than 7 kg undergoing an infra-umbilical surgery of expected duration of less than 1 hour. This strategy ensures the child's comfort and allows the procedure to be performed under optimal conditions for practitionner.
* The objective of this study is to review our practices and to evaluate the impact of the use of dexmedetomidine during spinal anesthesia of newborns and infants.

ELIGIBILITY:
Inclusion criteria:

* Newborns or Infants
* less than 7 kg
* Infra-umbilical surgery less than 1 hour
* Spinal anesthesia

Exclusion criteria:

* parental refusal
* Contraindication to spinal anaesthesia (coagulation disorder, ongoing sepsis, spinal malformation...).
* Contraindication to Dexmedetomidine (intracardiac conduction disorder, uncontrolled hemodynamic instability, alertness disorder)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All children weighing less than 7 kg undergoing an infra-umbilical surgery of expected duration of less than 1 hour
Sampling Method: Non-Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-11-28 (Estimated)

PRIMARY OUTCOMES:
duration of motor block | immediately after procedure in the recovery room
  Time at which the motor block is finished

CONTACTS AND LOCATIONS:
Overall Officials: Chrystelle SOLA, PH, Study Director — UH Montpellier
Locations (1):
- University Hospital, Montpellier, Hérault, France

IPD SHARING:
Plan to Share IPD: Undecided
NC